CLINICAL TRIAL: NCT00100035
Title: Polarity Therapy for Dementia Caregivers
Brief Title: Polarity Therapy for American Indian Caregivers of Dementia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001627-01A1 (NIH)
Record Dates: First submitted 2004-12-22; First posted 2004-12-23 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Stress; Depression; Anxiety
Keywords: Caregivers; Complementary Therapies
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Polarity therapy

SUMMARY:
The purpose of this study is to assess the effectiveness of polarity therapy (PT), a complementary and alternative medicine treatment, in American Indian caregivers living in the Pacific Northwest.

DETAILED DESCRIPTION:
The caregivers of people with dementia experience high levels of stress and are at particularly high risk for physical and mental illness. Although stress and illness are serious problems among American Indian caregivers in the Northwest, few studies have concentrated on this population. PT is a treatment that involves awareness of one's energy field and touch therapy; it has been shown to provide several physiological, biological, and psychological benefits. This study will determine whether PT is more effective than respite from caregiving in reducing stress, anxiety, and depression and improving health function and overall quality of life in American Indian caregivers.

Participants will be randomly assigned to receive either eight weekly sessions of PT or 3 hours of weekly respite from caregiving for 8 weeks. At the beginning of the study and at Weeks 4 and 8, participants will complete questionnaires and self-report scales on stress, anxiety, depression, and quality of life. In addition, heart rate variability and levels of cortisol will be measured at study entry and Weeks 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of a family member with dementia for at least 4 hours a day
* American Indian

Exclusion Criteria:

* Nerve disorders caused by diabetes
* Use of beta blockers

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Leslie E. Korn, PhD, MPH, Principal Investigator — Center for World Indigenous Studies
Locations (1):
- Center for World Indigenous Studies, Olympia, Washington, United States

REFERENCES:
- See also: Click here for more information about The Center for Traditional Medicine. — http://www.centerfortraditionalmedicine.org
- See also: Click here for more information on The Center for World Indigenous Studies. — http://www.cwis.org